CLINICAL TRIAL: NCT01938391
Title: Tissue Removal Assessment With Ultrasound of THe SFA and Popliteal (TRUTH Study)
Brief Title: Tissue Removal Assessment With Ultrasound of THe SFA and Popliteal
Acronym: TRUTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRUTH
Record Dates: First submitted 2013-03-12; First posted 2013-09-10 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Artery Disease; PAD; Claudication; Peripheral Vascular Disease; PVD
Keywords: Peripheral Artery Disease; PAD; Claudication; Peripheral Vascular Disease; PVD; Orbital Atherectomy; Balloon Angioplasty; Intravascular Ultrasound (IVUS)
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OAS + BA (Other): Cardiovascular Systems, Inc. Orbital Atherectomy System (OAS), is used prior to adjunctive balloon angioplasty (BA)
  Interventions: Device: Stealth 360°® OAS

INTERVENTIONS:
Device: Stealth 360°® OAS — Cardiovascular Systems, Inc. Orbital Atherectomy System (OAS) is used prior to adjunctive balloon angioplasty (BA)

SUMMARY:
IVUS imaging will be utilized to assess performance of the Sponsor's Orbital Atherectomy System (OAS) followed by adjunctive balloon angioplasty (BA) in patients who have symptomatic peripheral artery disease (PAD) occurring in the Superficial Femoral Artery (SFA), Popliteal (POP), and/or Tibioperoneal Trunk (TPT).

DETAILED DESCRIPTION:
This study is a prospective, single-arm (non-randomized), post-market study which will enroll up to 25 subjects. Intravascular Ultrasound (IVUS) imaging and angiography will be used to assess procedural outcomes in patients who have symptomatic peripheral artery disease who are treated with the Sponsor's OAS and adjunctive balloon angioplasty. An independent IVUS Core Lab will be used to provide adjudicated analyses for IVUS outcomes. In clinic follow-up visits will be performed at 2 weeks, 6 months and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age ≥ 18 years
* Subject is an acceptable candidate for percutaneous intervention using the Sponsor's OAS in accordance with its labeled indications and instructions for use
* Target lesion(s) located in a superficial femoral artery (SFA), popliteal (POP) or tibioperoneal trunk (TPT)
* Tight lesions (>70% stenosis)
* Lesions less than 110 mm in length
* Artery with the vessel < 6.5 mm in diameter
* Subject is willing and able to sign an approved informed consent form
* Subject is willing and able to attend follow-up visits

Exclusion Criteria:

* Uncontrolled allergy to nitinol, stainless-steel or other stent materials or to contrast agent
* Unable to take appropriate antiplatelet therapy
* Subject has no distal run-off
* Interventional treatment is intended for in-stent restenosis at the peripheral vascular site
* Subject has history of coagulopathy or hypercoagulable disorder, is undergoing hemodialysis or has impaired renal function (Cr > 2.5 mg/dl) at the time of treatment
* Female subject who is pregnant or nursing a child
* Intended interventional treatment includes planned laser, brachytherapy or atherectomy procedure other than the Sponsor's OAS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anvar Babaev, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
CSI has no plans to share IPD with other researchers

REFERENCES:
- [Result] Babaev A, Zavlunova S, Attubato MJ, Martinsen BJ, Mintz GS, Maehara A. Orbital Atherectomy Plaque Modification Assessment of the Femoropopliteal Artery Via Intravascular Ultrasound (TRUTH Study). Vasc Endovascular Surg. 2015 Oct;49(7):188-94. doi: 10.1177/1538574415607361. Epub 2015 Oct 20. PMID 26490645
- [Result] Krishnan P, Martinsen BJ, Tarricone A, Babaev A, Maehara A. Minimal Medial Injury After Orbital Atherectomy. J Endovasc Ther. 2017 Feb;24(1):167-168. doi: 10.1177/1526602816678033. Epub 2016 Nov 19. No abstract available. PMID 27864454

RESULTS

PARTICIPANT FLOW:
Groups:
- Stealth 360°® OAS: Cardiovascular Systems Inc.'s Orbital Atherectomy System (OAS), is used prior to adjunctive balloon angioplasty (BA)
  Stealth 360°® OAS: Cardiovascular Systems Inc. Orbital Atherectomy System (OAS) is used prior to adjunctive balloon angioplasty (BA)
Period: Baseline
Arm/Group | Stealth 360°® OAS
Started | 25
Completed | 25
Not Completed | 0
Period: 2 Week Follow up
Arm/Group | Stealth 360°® OAS
Started | 25
Completed | 25
Not Completed | 0
Period: 6 Month Follow up
Arm/Group | Stealth 360°® OAS
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: 12 Month Follow up
Arm/Group | Stealth 360°® OAS
Started | 24
Completed | 22
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Subjects with symptomatic peripheral artery disease
Arm/Group | Stealth 360°® OAS
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Number of treated lesions [Number; unit: lesions] | 29

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinically Driven Target Lesion Revascularization (TLR)
Description: A Kaplan-Meier analysis was performed to determine the percent probability that a study participant had a TLR at 6 months and at 12 months.
Time Frame: 6 months and 12 months
Measure: Number (95% Confidence Interval); unit: % probablity of clinically driven TLR
Arm/Group | Stealth 360°® OAS
Number analyzed (Participants) | 25
% probablity of clinically driven TLR
  TLR at 6 months | 4.0 [-3.7 to 11.7]
  TLR at 12 months | 8.2 [-2.7 to 19.0]

2. Primary Outcome: Mean Maximum Balloon Inflation Pressure
Description: Mean maximum balloon inflation pressure of balloons used pre-stent placement.
Time Frame: Index Procedure
Measure: Mean (Standard Deviation); unit: atm
Units Other Than Participants: balloons
Arm/Group | Stealth 360°® OAS
Number analyzed (Participants) | 25
Number analyzed (balloons) | 31
atm | 5.2 (1.2)

3. Primary Outcome: Rate of Procedural Angiographic Complications
Description: Percent of study participants with an Investigator reported procedural angiographic complication (flow limiting dissection, perforation, slow flow/no flow, distal embolization and recoil).
Time Frame: Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Stealth 360°® OAS
Number analyzed (Participants) | 25
Participants
  Flow limiting dissections (type D-F) | 0
  Perforations | 0
  Slow flow/no reflow | 0
  Distal embolization | 4
  Recoil | 0

4. Primary Outcome: Ankle-Brachial Index (ABI) Measurments
Description: The ankle-brachial index (ABI) is the ratio of the systolic blood pressure (SBP) measured at the ankle to that measured at the brachial (upper arm) artery. Normal range of ABI is 0.9 - 1.2. Values less than 0.9 suggests presence of peripheral artery disease (PAD). Values greater than 1.2 suggests of non-compressible vessel.
Time Frame: Baseline, 2 weeks, 6 months and 12 months
Population: At the time of this analysis 3 of the subjects did not have their ABI measured at baseline, 1 participant did not have their ABI measured at 2 weeks, 1 participant did not have their ABI measured at 6 months and 1 participant did not have their ABI measured at 12 months.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stealth 360°® OAS
Number analyzed (Participants) | 25
ratio
  ABI at Baseline: number analyzed (Participants) | 22
  ABI at Baseline | 0.74 (0.13)
  ABI at 2 weeks: number analyzed (Participants) | 24
  ABI at 2 weeks | 1.01 (0.10)
  ABI at 6 months: number analyzed (Participants) | 23
  ABI at 6 months | 0.96 (0.18)
  ABI at 12 months: number analyzed (Participants) | 21
  ABI at 12 months | 0.95 (0.15)

5. Primary Outcome: Rutherford Classification (RC)
Description: Rutherford Classification (RC) is a commonly used clinical grading system for describing peripheral arterial disease (PAD) on a scale of 0 to 6. RC 6 is the most severe form of PAD. The RC is assessed for each participant at baseline and at each follow-up visit.
  RC classification is as follows:
  RC 0: Asymptomatic, no hemodynamically significant occlusive disease RC 1-3: Mild to Severe Claudication, limitation with ordinary physical activities, patient is comfortable at rest RC 4-5: Ischemic rest pain, minor tissue loss, non healing ulcer, focal gangrene RC 6: Major tissue loss, functional foot no longer salvageable
Time Frame: Baseline, 2 weeks, 6 month and 12 month
Population: At the time of analysis for the 6 month visit 1 participant missed their follow up visit. At the time of analysis for the 12 month visit, 22 participants completed the 12 month follow up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Stealth 360°® OAS
Number analyzed (Participants) | 25
Participants
  RC 0 at baseline | 0
  RC 0 at 2 weeks | 24
  RC 0 at 6 month: number analyzed (Participants) | 24
  RC 0 at 6 month | 19
  RC 0 at 12 month: number analyzed (Participants) | 22
  RC 0 at 12 month | 13
  RC 1 at baseline | 0
  RC 1 at 2 weeks | 1
  RC 1 at 6 month: number analyzed (Participants) | 24
  RC 1 at 6 month | 2
  RC 1 at 12 months: number analyzed (Participants) | 22
  RC 1 at 12 months | 8
  RC 2 at baseline | 0
  RC 2 at 2 weeks | 0
  RC 2 at 6 month: number analyzed (Participants) | 24
  RC 2 at 6 month | 0
  RC 2 at 12 months: number analyzed (Participants) | 22
  RC 2 at 12 months | 1
  RC 3 at baseline | 25
  RC 3 at 2 weeks | 0
  RC 3 at 6 month: number analyzed (Participants) | 24
  RC 3 at 6 month | 3
  RC 3 at 12 months: number analyzed (Participants) | 22
  RC 3 at 12 months | 0

6. Primary Outcome: Stent Usage at the Time of the Index Procedure
Description: Number of lesions with a stent placed during the index procedure.
Time Frame: Index Procedure
Population: Number of stents placed is based on number of lesions treated in the total subject population of 25. The total number of lesions treated were 29 and of those 29 lesions, 17 had a stent placed.
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Stealth 360°® OAS
Number analyzed (Participants) | 25
Number analyzed (Lesions) | 29
Lesions | 17

7. Primary Outcome: Percent (%) Area Stenosis
Description: Percentage (%) of area stenosis as assessed by the intravascular ultrasound (IVUS) Core Lab. Percentage of area stenosis was calculated as 1 - (minimum lumen area / reference lumen area).
Time Frame: Index Procedure (pre-procedure, post-OAS treatment and post-balloon treatment)
Population: At the time of analysis 24 of 29 lesions in 25 participants could be assess by the IVUS Core Lab.
Measure: Median (Inter-Quartile Range); unit: percent area stenosis
Units Other Than Participants: lesions
Arm/Group | Stealth 360°® OAS
Number analyzed (Participants) | 25
Number analyzed (lesions) | 24
percent area stenosis
  Pre-procedure, Area Stenosis (%) | 76.9 [61.3 to 80.5]
  Post-OAS treatment, Area Stenosis (%) | 63.8 [57.6 to 76.7]
  Post-Balloon treatment, Area Stenosis (%) | 43.0 [27.3 to 56.4]

ADVERSE EVENTS:
Time Frame: AEs were collected during the index-procedure through 12 months of follow up.
Arm/Group | Stealth 360°® OAS
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stealth 360°® OAS (N=25)
Bleeding, access site (Injury, poisoning and procedural complications) | 1 (1)
Distal Embolization (Injury, poisoning and procedural complications) | 4 (4)
Dissection (Injury, poisoning and procedural complications) | 2 (2) — All dissections were non-flow limiting
Chest Pain (Cardiac disorders) | 1 (1)
Worsening of PAD (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stealth 360°® OAS (N=25)
Dissection (Injury, poisoning and procedural complications) | 10 (10) — All dissections were non-flow limiting
Worsening of PAD (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
TRUTH was a single center, non-randomized trial that enrolled a small number of subjects (25).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less